CLINICAL TRIAL: NCT02848170
Title: An Exploratory Study of CS-3150 to Evaluate the Relation Between Antihypertensive Effect and Baseline Factors Compared to Olmesartan Medoxomil in Patients With Essential Hypertension
Brief Title: Study of CS-3150 Compared to Olmesartan in Patients With Essential Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CS3150-A-J303
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2017-05

CONDITIONS: Essential Hypertension
Keywords: essential hypertension; mineralocorticoid receptor antagonist; Developmental Phase III
MeSH Terms: conditions — Essential Hypertension | interventions — esaxerenone; Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CS-3150 (Experimental): CS-3150 2.5 to 5mg, orally, once daily after breakfast for 12 weeks
  Interventions: Drug: CS-3150
- olmesartan medoxomil (Active Comparator): olmesartan medoxomil 10 to 20 mg, orally, once daily after breakfast for 12 weeks
  Interventions: Drug: olmesartan medoxomil

INTERVENTIONS:
Drug: CS-3150 — CS-3150 2.5mg, oral
  Arms: CS-3150
Drug: olmesartan medoxomil — olmesartan medoxomil 10 mg, oral
  Other Names: Benicar
  Arms: olmesartan medoxomil

SUMMARY:
Phase 3 study to examine the relation between antihypertensive effect and baseline factors exploratively, compared to olmesartan medoxomil in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 20 years or older at informed consent
* Subjects with essential hypertension during run-in period (mean 24 hour systolic blood pressure SBP ≥ 130 and diastolic blood pressure DBP ≥ 80 mmHg and Sitting systolic blood pressure (SBP) ≥ 140 mmHg and < 180 mmHg, Sitting diastolic blood pressure (DBP) ≥ 90 mmHg and < 110 mmHg)

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* Diabetes mellitus with albuminuria
* Serum potassium level < 3.5 or ≥ 5.1 milliequivalent (mEq)/L
* Reversed day-night life cycle including overnight workers
* estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m^2.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24 hr blood pressure | baseline to end of Week 12
  Relationship between the change from baseline in 24 hr blood pressure (systolic, diastolic, and average blood pressure) and baseline factors frpm baseline to end of Week 12

SECONDARY OUTCOMES:
Change from baseline in morning, evening, and night blood pressure. | baseline to week 12
  Relationship between the change from baseline in morning, evening, and night blood pressure (systolic, diastolic, and average blood pressure) and baseline factors.
Change from baseline in sitting blood pressure | baseline to week 12
  Relationship between the change from baseline in sitting blood pressure (systolic, diastolic, and average blood pressure) and baseline factors.
Time course of 24 hr blood pressure and sitting blood pressure | week 12
  Time course of 24 hr blood pressure and sitting blood pressure (systolic, diastolic, and average blood pressure)
Proportion of patients achieving 24 hr and sitting blood pressure control | week 12
  Proportion of patients achieving 24 hr and sitting blood pressure control

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/